CLINICAL TRIAL: NCT02307006
Title: IDC 56: A Randomized Double-blinded Study Comparing Ceftaroline to Standard of Care Therapy With Cefazolin and Vancomycin as Surgical Prophylaxis for High Risk Orthopedic and Cardiac Surgeries
Brief Title: The Use of Ceftaroline as Surgical Prophylaxis in Surgery With Risk of MRSA Infection
Acronym: PREVTAROLINE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cincinnati (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, George Smulian, Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IDC 56 / IIT-USA-000585/
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Ceftaroline; Cefazolin; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ceftaroline (Experimental): Experimental comparator for surgical peri-operative prophylaxis for procedures at increased risk if MRSA infection
  Interventions: Drug: Ceftaroline
- Cefazolin / Vancomycin (Active Comparator): Standard of care comparator for surgical peri-operative prophylaxis for procedures at increased risk if MRSA infection
  Interventions: Drug: Cefazolin / Vancomycin

INTERVENTIONS:
Drug: Ceftaroline — Surgical prophylaxis
  Other Names: Teflaro
  Arms: Ceftaroline
Drug: Cefazolin / Vancomycin — Standard of care surgical prophylaxis
  Other Names: Ancef; Vancin
  Arms: Cefazolin / Vancomycin

SUMMARY:
The study is a randomized double-blinded study comparing ceftaroline to standard of care therapy with cefazolin and vancomycin as surgical prophylaxis for high risk orthopedic and cardiac surgeries. Study participants will be enrolled from those undergoing cardiothoracic surgery involving sternotomy and those undergoing prosthetic joint replacement of either hip or knee. Consenting patients will be randomized 2:1 to receive either ceftaroline or cefazolin/vancomycin. This study will be blinded by the use of placebo vancomycin infusions and placebo cephalosporin infusions. The primary end point will be the development of a surgical site infection within 30 days of surgery.

DETAILED DESCRIPTION:
The study is a randomized double-blinded study comparing ceftaroline to standard of care therapy with cefazolin and vancomycin as surgical prophylaxis for high risk orthopedic and cardiac surgeries. Study participants will be enrolled from those undergoing cardiothoracic surgery involving sternotomy and those undergoing prosthetic joint replacement of either hip or knee. Consenting patients will be randomized 2:1 to receive either ceftaroline or cefazolin/vancomycin. This study will be blinded by the use of placebo vancomycin infusions and placebo cephalosporin infusions. Study participants will be enrolled from 2 populations of patients; those undergoing cardiothoracic surgery with sternotomy and those undergoing prosthetic joint replacement of either hip or knee.

Subjects will be identified by the primary surgical service. Adult subjects 18 years and older will be notified of the study and if agreeable will be interviewed by a study coordinator who will explain the study and study procedures and determine eligibility. Informed consent will be obtained from potential participants. Enrollment and consent may be obtained up to seven days prior to surgery.

Consented participants will have a detailed history performed with particular reference to prior surgical infections, risk factors such as diabetes, smoking, prior skin infections and obesity. Participants will undergo a physical examination. Patients will be assessed for nares colonization with methicillin-resistant Staphylococcus aureus (MRSA) as per the primary surgeon's standard procedure. Patients identified as positive for MRSA colonization will be decolonized with mupirocin. Female participants will have a serum beta-human chorionic gonadotrophin (HCG) assay performed to exclude pregnancy.

Consented participants will be randomized 2:1 to receive either ceftaroline or cefazolin/vancomycin, the current regimen for high risk individuals. Randomization will be performed by a blinded individual using a randomization program. Within each group, participants will be allocated in the 2:1 ratio.

On the day of surgery, all patients will be evaluated for changes in medical history, vital signs recorded and bilateral nares swabs obtained for Staphylococcal screening for both MRSA and methicillin-sensitive Staphylococcus aureus (MSSA) carriage. All patients will receive pre-operative toweling of the operative site with chlorhexidine, and a surgical skin preparation of chlorhexidine/alcohol (Duraprep).

Consented participants will receive two blinded infusions. Study infusions will be prepared by an unblinded pharmacist to match the active medications. Placebo and study medication will be matched in volume and appearance. Dosing of vancomycin and cefazolin will be weight based up to 120 kg at 15 mg/kg and 25 mg/kg respectively. ceftaroline will be administered at a dose of 600 mg in individuals with estimated creatinine clearance of greater than 50 ml/min and 400 mg for those with creatinine clearance rates of 30-50 ml/min. Vancomycin or placebo1 will be started 120 minutes prior to incision and completed within 60 minutes prior to surgery. The cefazolin or ceftaroline will be started 60 minutes before surgery and completed 30 minutes prior to incision. Each participant will thus receive 2 infusions at T-120 and T-60 minutes from time of skin incision.

Patients will be redosed with antibiotics between 1.5 to 2 half-lives (cefazolin or ceftaroline at 4hrs hours post skin incision and vancomycin/placebo 1 at 12 hrs) in prolonged procedures. One post-operative dose of of cefazolin/ceftraroline will be given in the recovery room 4 hours after skin incision for those patients who were not redosed during the procedure for orthopedic procedures and 2 doses will be administered for cardiothoracic procedures.

Pharmacokinetic substudy:

Because of the variation in the pharmacokinetics previously identified for patients undergoing extracorporeal circulation, we will perform a pharmacokinetic analysis on a subset of 50 patients in the cardiac surgery arm of the study to allow data on at least 30 patient receiving ceftaroline. Plasma samples will be collected at the start of infusion (time = 0, Sample #1), end of infusion (time = 30 minutes, Sample #2), 15 minutes post infusion (Sample #3), at the time of skin incision (Sample #4) at commencement of cardiopulmonary bypass (CPB) (Sample # 5), at completion of CPB (Sample # 6) and at the time of skin closure (Sample #7). Samples will be analyzed by high pressure liquid chromatography (HPLC) to determine ceftaroline levels using known plasma standards with appropriate quality controls.

Patients will undergo a wound inspection by study personnel prior to discharge from hospital. Microbiological cultures will be obtained from all surgical site infections. All isolates will be reported out. Patients will be interviewed and examined at day 30 for the presence of evidence of surgical site infection at any operative site. Subjects will be questioned with regard to the presence of fever, redness or drainage or other manifestations of infection. Physical examination findings by the surgical team at prior post-operative visits will be reviewed and correlated with the data obtained from the subject. The primary end point will be the development of a surgical site infection within 30 days of surgery.

30 day surgical site infection rates at either the primary surgical site or any remote surgical site (e.g. vein donor site for CABG procedures) will be used as the principal outcome measure. Surgical site infections will be characterized as superficial (above the fascia) or complex (deep (extending below the fascia) and organ involving), Secondary endpoints recorded will include (i) other infections, viz. pulmonary, UTI, line related); (ii) Drug related, viz., rash, itching; and (iii) nausea, vomiting and (iiii) return to OR.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Age - 18 years and older
* Patients undergoing either hip or knee arthroplasty or cardiac surgery with sternotomy
* Body mass index (BMI) between 18 and 30 kg/m2 inclusive.
* Female subjects must have a negative serum pregnancy test and be using appropriate contraception.

Exclusion Criteria:

* Pregnancy
* Hypersensitivity or allergic reaction to any β-lactam antibiotic or vancomycin.
* Presence of cardiovascular shock,
* Receipt of chronic concomitant systemic corticosteroids, 40 mg of prednisone equivalent;
* Severe renal impairment (i.e. Creatinine clearance ≤ 30 mL/min);
* Significant hepatic impairment (i.e. known acute viral hepatitis, aspartate aminotransferase or alanine aminotransferase concentration 10-fold the upper limit of normal (ULN) or total bilirubin 3-fold the ULN or manifestations of end-stage liver disease, such as ascites or hepatic encephalopathy),
* Hematological impairment with current or anticipated neutropenia with less than 500 neutrophils/mm3 or thrombocytopenia with platelet count of 60 000 cells/mm3
* HIV infection which at the time of screening meets 2008 CDC criteria for AIDS.
* Patients undergoing revision surgery for infected prosthetic joint replacement.
* Body mass index (BMI) less than 18 or greater than 30 kg/m2.
* Concurrent antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection | 30 days
  Surgical site infection rates at either the primary surgical site or any remote surgical site

SECONDARY OUTCOMES:
Other infection | 30 days
  Other infections, viz. pulmonary, UTI, line related
Drug intolerance | 30 days
  Drug related, viz., rash, itching, nausea, vomiting
Repeat surgery | 30 days
  Return to OR

CONTACTS AND LOCATIONS:
Overall Officials: Alan G Smulian, M.B.B.Ch., Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - West Chester Hospital, West Chester, Ohio